CLINICAL TRIAL: NCT04648748
Title: Normative Data of Hand Grip Strength in Healthy Adult Pakistani Population
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/19/1005 Danish Hassan
Record Dates: First submitted 2020-11-15; First posted 2020-12-01 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Health, Subjective
Keywords: Hand Grip Strength; Normative Data; Healthy Adults

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Normative data values of handgrip strength not only describes hand normality but is also used as an objective assessor of upper extremities damages for Occupational Therapy and Physical Therapy interventions. Published normative data of different populations are widely available and can be used as reference. It is evident from different researches that various anthropometric variables such as age, gender, ethnicity, nutritional status, shoulder circumference & Body Mass Index(BMI), type of occupation and hand dominance of any population influence the hand muscles grip strength. Whereas, some literature shows disparity over the correlation between hand grip strength and BMI, several researchers claiming a positive relationship between BMI and grip strength in all ages of both genders, while other indicates no relationship.

Approximately 3000 volunteers will be recruited from the staff, medical students, and visitors of different medical college & universities of Lahore. Subjects will be excluded if they had a history of upper-limb injury or deformity, or related health conditions. Socioeconomic background, general health, and lifestyle of the subjects will be assessed using a standard questionnaire. Weight, height & APM thickness will be measured prior to testing. Correlation between Hand Grip Strength and age, weight, height, body mass index (BMI), and Adductor Polices Muscle Thickness (APMT) will be measured. Multiple linear regression analysis will be used to adjust for the effects of other variables and to identify those independently associated with Hand grip strength. All the analysis will be carried out on SPSS v 25.

DETAILED DESCRIPTION:
In the last 20 years, a number of scientific publications from around the world point to hospital malnutrition as a direct cause for higher morbidity (slower wound healing; higher hospital infection rates; longer stay, especially among intensive care patients; higher readmission rates) and mortality. The obvious impact of such a scenario include avoidable deaths, additional costs for the social security system, and the social onus related to loss of working days.

A wide variety of methods are available for nutritional evaluation. Not with standing, none of these can currently be considered as a ''gold-standard'' for diagnosing hospital malnutrition. Available methods include anthropometry, the creatinine height index, albumin, pre-albumin, immuno competence evaluation, cholesterol, and the prognostic nutritional index, among others. However, none of these methods provides a functional evaluation of malnutrition. SGA is a well-accepted method of nutritional assessment that addresses functional status as a complement of its medical history, but it was not developed to be used to evaluate responsiveness, and so, its rating are not expected to show any modification after nutritional interventions in short periods of time.

There is evidence that muscular function is altered and muscular strength diminished, in the presence of malnutrition. According to Jeejeebhoy, malnutrition-related muscular function alterations appear before changes in anthropometric and laboratory parameters. Nevertheless, methods for evaluating muscular strength during nutritional evaluation are still scarce. The earliest nutritional alterations occur within muscle cells, and have an effect on muscle cell function. Measuring muscular strength may therefore provide a sensitive method for nutritional evaluation. Muscular loss is inevitable during malnutrition, and if untreated, may become progressive. Therefore, in addition to their ability to detect early alterations related to malnutrition, muscular function tests could also prove useful for evaluating nutritional recovery, underscoring the importance of such evaluation in this context.

Recent studies have demonstrated the validity of using hand dynamometers as a method for nutritional evaluation, given that this is a simple, fast, useful, inexpensive, and efficacious test for muscular function. Knowledge of reference values in a healthy population would allow a functional muscle evaluation not only in hospital and research settings, but also in population-based studies. The aim of the study is to determine reference values and associated factors for hand grip strength in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects as measured on Subjective Global Assessment Form

Exclusion Criteria:

* History/o upper limb surgery, deformity or related health condition
* No previous history pf participation in gym activities for last 06 months

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be recruited from the staff, medical students, and visitors of different medical college & universities of Lahore. Subjects will be excluded if they had a history of upper-limb injury or deformity, or related health conditions. Socioeconomic background, general health, and lifestyle of the subjects will be assessed using a standard questionnaire. Weight, height & APM thickness will be measured prior to testing.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength | 3 Weeks
  Hand grip strength can be quantified by measuring the amount of static force that the hand can squeeze around a dynamometer. The force has most commonly been measured in kilograms and pounds, but also in millilitres of mercury and in Newtons

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lam NW, Goh HT, Kamaruzzaman SB, Chin AV, Poi PJ, Tan MP. Normative data for hand grip strength and key pinch strength, stratified by age and gender for a multiethnic Asian population. Singapore Med J. 2016 Oct;57(10):578-584. doi: 10.11622/smedj.2015164. Epub 2015 Nov 13. PMID 26768064
- [Background] Lim SH, Kim YH, Lee JS. Normative Data on Grip Strength in a Population-Based Study with Adjusting Confounding Factors: Sixth Korea National Health and Nutrition Examination Survey (2014-2015). Int J Environ Res Public Health. 2019 Jun 25;16(12):2235. doi: 10.3390/ijerph16122235. PMID 31242569
- [Background] Angst F, Drerup S, Werle S, Herren DB, Simmen BR, Goldhahn J. Prediction of grip and key pinch strength in 978 healthy subjects. BMC Musculoskelet Disord. 2010 May 19;11:94. doi: 10.1186/1471-2474-11-94. PMID 20482832
- [Background] Dodds RM, Syddall HE, Cooper R, Benzeval M, Deary IJ, Dennison EM, Der G, Gale CR, Inskip HM, Jagger C, Kirkwood TB, Lawlor DA, Robinson SM, Starr JM, Steptoe A, Tilling K, Kuh D, Cooper C, Sayer AA. Grip strength across the life course: normative data from twelve British studies. PLoS One. 2014 Dec 4;9(12):e113637. doi: 10.1371/journal.pone.0113637. eCollection 2014. PMID 25474696
- [Background] Shim JH, Roh SY, Kim JS, Lee DC, Ki SH, Yang JW, Jeon MK, Lee SM. Normative measurements of grip and pinch strengths of 21st century korean population. Arch Plast Surg. 2013 Jan;40(1):52-6. doi: 10.5999/aps.2013.40.1.52. Epub 2013 Jan 14. PMID 23362480